CLINICAL TRIAL: NCT06495047
Title: Assessment of Optimal Inhaler Therapy Strategies in the Management of Acute Exacerbations of COPD (AECOPDs) Using Oscillometry: A Cross-Sectional Study
Brief Title: Assessing Optimal Inhaler Strategies During Acute Exacerbations of COPD (AECOPDs) Using Oscillometry
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: MEI/MES I&P Program (McGill University, Thorasys Inc.) (Unknown)
Responsible Party: Principal Investigator, Bryan Ross, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2024-10445
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: COPD; COPD Exacerbation Acute
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD cohort: Males and females aged 40 or greater with any severity of airflow obstruction (GOLD 1-4) who are currently experiencing and receiving treatment for a physician-diagnosed acute exacerbation (AECOPD) with both long-acting and short-acting bronchodilators prescribed by the treating team.
  Interventions: Drug: Long-acting bronchodilator therapy (LABD); Drug: Short-acting bronchodilator therapy (SABD)

INTERVENTIONS:
Drug: Long-acting bronchodilator therapy (LABD) — Long-acting inhaler therapy
Drug: Short-acting bronchodilator therapy (SABD) — Short-acting inhaler therapy

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a persistent lung disease that makes it very difficult to breathe. The airways and the normally 'spongy' lungs themselves are affected. The main treatment is puffers, some which are long-acting (to control persistent symptoms) and some which are short-acting ('rescue' puffers when suddenly feeling short-of-breath). Beyond persisting breathlessness at rest, people with COPD can also experience dangerous "lung-attacks" which can require urgent care visits or even hospitalization for treatment. Amazingly, although COPD is the third leading cause of death worldwide, and COPD lung-attacks are a leading cause of hospitalization in Canada, investigators are still unsure which combination of puffers is most effective at treating lung-attacks.

The main objective is to determine which puffer treatment combination (just short-acting, or both short-acting and long-acting) best opens up the lungs to airflow during COPD lung-attacks.

A test called oscillometry, which requires only quiet breathing and is so safe that it is regularly used in children, toddlers and even infants, will be used to measure lung function changes. All eligible people with COPD receiving urgent lung-attack treatment who agree to participate will perform three rounds of oscillometry: before any puffers, after only short-acting puffers, and finally after long-acting puffers are also added on. Any potential evidence of side effects will be collected from the chart. Oscillometry tests will be compared to see which puffer strategy best improves flow in the airways.

Part of the reason why this has not been well-studied so far is that the standard breathing test, spirometry, requires multiple rounds of forceful breathing which is very difficult, even distressing, for many people with COPD (at rest, let alone during a lung-attack). No studies have ever properly studied which puffer strategy is most effective for lung-attacks. The investigators have experience and expertise with oscillometry, the most appropriate test in this setting, to answer this pressing question.

This research addresses an important treatment knowledge gap for this very common lung disease. These results could influence how patients with COPD around the world are treated during lung-attacks so that they can breathe better, sooner.

DETAILED DESCRIPTION:
Three sets of carefully timed oscillometry and dyspnea score measurements will be performed: 1) at "baseline", before the participant receives their scheduled dose of LABD and roughly 4 hours following a scheduled dose of SABD; 2) between 15-20 min after having received their next scheduled dose of SABD and just preceding their next scheduled dose of LABD (SABD only); and 3) after having received the scheduled dose of LABD and between 25-35min of the most recent SABD administration (LABD + SABD), such that there is overlap in the time window of SABD and LABD onset at the time of the third set of testing.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥ 40, who are former/current smokers with a ≥10 pack-year smoking history.
2. COPD previously confirmed by spirometry (FEV1/FVC < 0.7) of any severity (GOLD 1-4).
3. Currently experiencing and receiving treatment for a physician-diagnosed AECOPD with both long-acting and short-acting bronchodilators prescribed by their treating team.
4. Ability to participate without supplemental oxygen during the oscillometry tests.
5. Ability to provide informed consent.

Exclusion Criteria:

1. No COPD diagnosis.
2. AECOPD is not the principal cause of urgent care visit, emergency department visit, or hospitalization.
3. Treatment strategy in which LABDs were held by the treating medical team (SABD-only approach).
4. Participant already performed spirometry on the same day of testing.
5. Inability to provide informed consent.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with COPD diagnosed with and receiving treatment for an acute exacerbation (AECOPD) who are being treated with both short-acting and long-acting bronchodilator therapies. Convenience sampling approach.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-11-19 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reactance-volume loop area (AXV) | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Parameter collected by intra-breath (within-breath) oscillometry. The area within the reactance-volume curve, during tidal breathing.
Mean inspiratory minus expiratory respiratory system reactance (mean ∆Xrs) | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Parameter collected by intra-breath (within-breath) oscillometry. The reactance during inspiration, minus the reactance during expiration, during tidal breathing.

SECONDARY OUTCOMES:
Visual analog scale (VAS) Dyspnea Score | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Validated visual representation of shortness of breath.
Resistance at 5 Hz (R5) | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Parameter collected by spectral oscillometry. The resistance as measured by oscillometry at 5 Hz.
Reactance at 5 Hz (X5) | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Parameter collected by spectral oscillometry. The reactance as measured by oscillometry at 5 Hz.
Frequency Dependence of Resistance (R5-20) | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Parameter collected by spectral oscillometry. The resistance as measured by oscillometry at a range from 5 Hz to 20 Hz.
Reactance Area (Ax) | 1) At baseline (before bronchodilators); 2) 15-20 minutes after SABD but before LABD; and 3) after SABD and LABD (25-35 minutes following SABD).
  Parameter collected by spectral oscillometry. The area under the reactance curve.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Due to data privacy regulations, individual participant data collected during this study is not publicly accessible. However, access to anonymized data may be granted upon evaluation by the trial management group. Additional documents will also be available upon inquiry. All requests should be directed to the corresponding author (BAR).